CLINICAL TRIAL: NCT05310487
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics of 162 With a Single Ascending Dose in Healthy Adult Subjects
Brief Title: Phase 1 Study of 162, a Novel Neutralizing Antibody Targeting Hepatitis B Surface Antigen, in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yangshengtang Co., Ltd (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YST-162-101
Record Dates: First submitted 2022-03-23; First posted 2022-04-05 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-07

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 162 (Experimental): The dose-escalation stage will be conducted sequentially at 5 dose levels, which are 100 mg in the pre-test, and 200 mg, 400 mg, 800 mg and 1200 mg in the formal test. Two healthy adult subjects will be enrolled at 100 mg dose level and all given 162. At the start of each level with the exception of 100 mg level which there are only two subjects, two sentinel subjects will be randomized 1:1 to 162 or placebo. The remaining subjects will be randomized 5:1 to receive a single ascending dose of 162 or placebo.
  Interventions: Biological: 162
- placebo (Placebo Comparator): At the start of each level with the exception of 100 mg level which there are only two subjects, two sentinel subjects will be randomized 1:1 to 162 or placebo. The remaining subjects will be randomized 5:1 to receive a single ascending dose of 162 or placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: 162 — The investigational product 162 is a novel neutralizing antibody targeting HBsAg, for the treatment of patients with chronic hepatitis B
  Arms: 162
Other: Placebo — an intervention that appearance is the same as 162, but contains no active ingredients
  Arms: placebo

SUMMARY:
This is the first in human study of 162, and the primary objective is to evaluate the safety and tolerability of 162 with a single ascending dose in healthy adult subjects.

The dose-escalation stage will be conducted sequentially at 5 dose levels, which are 100 mg in the pre-test, and 200 mg, 400 mg, 800 mg and 1200 mg in the formal test.

Two healthy adult subjects will be enrolled at 100 mg dose level and all given 162. Eight healthy adult subjects will be enrolled at each remaining dose levels (200 mg, 400 mg, 800 mg and 1200 mg), respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the study, be able to understand the requirements of a clinical study, and sign informed consent form.
2. Aged ≥ 18 and ≤ 55 years older, male and female.
3. Body weight ≥ 50 kg for male, body weight ≥ 45 kg for female, and body mass index (BMI) scores between ≥ 18 kg/m2 and ≤ 32.0 kg/m2.
4. Vital signs, physical examination, laboratory tests and 12-lead ECG, etc. within normal limits; or, with no clinically significant abnormalities as determined by the investigator.
5. A male participant must agree to use adequate contraception from screening through at least 12 weeks after the last dose of investigational product or placebo. Refer to Section 5.5 for more information on highly effective methods of contraception.
6. Women of childbearing potential must have a negative pregnancy test prior to the dosing administration, and agree to use adequate contraception from screening through at least 12 weeks after the last dose of investigational product or placebo. A female participant of non-childbearing potential will have had at least 12 continuous months of natural (spontaneous) amenorrhoea, follicle stimulating hormone (FSH) level > 40 mIU/mL at screening, and an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms); or have had surgical bilateral oophorectomy, hysterectomy or tubal ligation beyond 6 weeks prior to screening. Refer to Section 5.5 for more information on highly effective methods of contraception

Exclusion Criteria:

1. History of anaphylaxis or clinically significant drug allergy or drug allergy witnessed in previous studies with experimental drugs, or allergy to the active ingredients or excipients of the investigational product.
2. History of allergic reactions to monoclonal antibodies or antibody fragments.
3. History or presence of infectious or non-infectious liver disease, including but not limited to a history of alcoholic liver disease, non-alcoholic steatohepatitis, drug or autoimmune liver disease.
4. History or presence of immune-mediated diseases, including but not limited to idiopathic thrombocytopenic purpura, systemic lupus erythematosus, rheumatoid arthritis.
5. History or presence of any chronic infectious condition, including but not limited to tuberculosis or parasitic infections.
6. History of allogenic transplantation of organs, bone marrow or stem cell.
7. Active infection, or screening for infectious disease during the screening period (HBsAg, hepatitis C virus antibody [HCV-Ab], human immunodeficiency virus antibody [HIV-Ab], or syphilis antibody [TP-Ab]) is positive.
8. QTcF >450 msec on 3 consecutive ECG recordings conducted at screening or baseline.
9. Alanine transaminase (ALT) > 1.2 × ULN, aspartate aminotransferase (AST) > 1.2 × ULN or total bilirubin > 1.2 × ULN.
10. Any other concomitant disease, condition or treatment that could interfere with the conduct of the study or that would, in the opinion of the Investigator or Sponsor, pose an unacceptable risk to the subject in the study or interfere with the interpretation of study data.
11. Took any prescription drugs or over-the-counter drugs within 2 weeks prior to investigational product or placebo administration, or took any drugs within 5 half-lives at the time of investigational product or placebo administration (whichever is longer), but vitamins, supplements and topical corticosteroids will be permitted within 2 weeks prior to investigational product or placebo administration; or, took any herbal medicines within 30 days before investigational product or placebo administration.
12. Those who have received live or attenuated vaccines (e.g., measles, mumps, rubella, varicella, yellow fever, rabies, BCG, typhoid vaccine, etc.) within 4 weeks before screening, or any covid-19 vaccine within 2 weeks before screening.
13. Those who donated plasma within 7 days prior to the dosing administration or donated or lost blood 500 mL or more within 8 weeks prior to the dosing administration, or plan to donate during the study or within 8 weeks after the end of the study.
14. Those who underwent surgery within 4 weeks before screening, or plan to undergo surgery during the study.
15. Those who are participating in other clinical studies, or currently not participating in a study and have been dosed in another clinical study in the past 4 weeks.
16. Pregnant or lactating women.
17. Those who are determined disqualified to join clinical studies by investigator for other causes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Day 1-Day 28
  incidence and severity of adverse events after the administrtion of 162 or placebo

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Day 1-Day 28
  Maximum concentration of 162 in blood after administration
Area under the plasma concentration versus time curve from time 0 to the last test time(AUC last) | Day 1-Day 28
  Area under the plasma concentration of 162 versus time curve from time 0 to the last test time
Area under the plasma concentration versus time curve from time 0 to infinity time(AUC 0-∞) | Day 1-Day 28
  Area under the plasma concentration of 162 versus time curve from time 0 to infinity time
Half life (t1/2) | Day 1-Day 28
  The elimination half-life time of 162 in blood
Clearance (Cl) | Day 1-Day 28
  Clearance of 162 in blood
Apparent volume of distribution (Vd) | Day 1-Day 28
  The apparent volume of distribution of 162 in vitro
Immunogenicity | Day 1-Day 28
  To evaluate the level of anti-drug antibody (ADA) produced by the subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No